CLINICAL TRIAL: NCT01499784
Title: Can Urinary Incontinence be Treated in an In-patient Rehabilitation Setting?
Brief Title: Urinary Incontinence in an Inpatient Rehab Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Deutsch (Other)
Collaborators: Shirley Ryan AbilityLab (Other)
Responsible Party: Sponsor-Investigator, Anne Deutsch, Principal Investigator, Shirley Ryan AbilityLab
Organization: Shirley Ryan AbilityLab (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 61418
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pelvic Floor muscle Training (Experimental): educational class for behavioral modification and group exercise class for pelvic floor muscle training
  Interventions: Behavioral: pelvic floor muscle training

INTERVENTIONS:
Behavioral: pelvic floor muscle training — behavioral modification and pelvic floor muscle training

SUMMARY:
Urinary incontinence (UI) is a very common condition in women, with estimates of prevalence varying from 10% to 40% in most studies and showing a gradual increase with age. UI is a serious medical problem that can lead to urinary tract infections, low back pain, respiratory disorders, pressure sores, and an increased risk of falls. It also leads to social problems, creating embarrassment and negative self-perception for those who suffer from it. Women with urinary incontinence find themselves isolated and relatively inactive. A wide range of treatments has been used in the management of women's UI, including conservative interventions, pharmaceutical intervention, and surgery. A Cochrane Review from 2008 stated that pelvic floor muscle training (PFMT) is better than no treatment for UI and supports the recommendation that PFMT should be the first treatment line in conservative management programs for women with UI. Recently, there have been a few articles published that looked at the effectiveness of treating UI in a group-like setting with both behavioral modifications and pelvic floor exercises. One study was able to prove that group training of behavioral modification helped to reduce UI severity, increase pelvic floor strength, and reduce voiding frequency when compared to a control group.

All of the studies cited were performed in community-dwelling persons with out-patient services and interventions. Dr. Fitzgerald and her colleagues from The Rehabilitation Institute of Chicago (RIC) were able to confirm in a poster presentation that many patients admitted to an inpatient rehabilitation facility do have UI. In 2005, out of 403,697 Medicare beneficiaries admitted to a rehab hospital, 24% were incontinent. These studies were able to illustrate that UI affects all diagnoses. UI was shown to make a significant contribution to patient outcomes independent of functional status at admission. It is also a large determinant of discharge destination. In the United Kingdom in 2004, 62% of incontinent stroke patients were discharged to a sub acute home with only 5% placement for continent stroke survivors. Another study determined that urinary incontinence after having a stroke predicted a higher likelihood of an adverse outcome when controlled for age, type of stroke, and length of hospital stay. May, et. al., was able to state while in an acute rehab setting that patients with spinal cord injuries ranked bowel and bladder care, along with skin care, as most important in an education class with 12 different topics. This shows that patients find bladder function a large priority in their care, even in an in-patient setting. In the poster presentation mentioned above, many patients with UI in an acute care rehab setting do not improve Functional Independence Measure (FIM) status from admission to discharge. Currently there is no research available for the treatment of UI in an acute care rehab hospital, though it has been shown to be an issue with many of those admitted. So the question arises, "Would addressing urinary incontinence with physical therapy interventions and behavioral modifications improve incontinence in this population during the acute rehab stage?"

DETAILED DESCRIPTION:
This project will look at the possibility of treating in-patients with UI at RIC while in the acute rehab hospital setting to determine what positive outcomes are possible. Subjects will be provided both individual and group sessions to help educate and treat those suffering with UI. Subjects would participate in a weekly educational class of lecture and video and then perform both pelvic floor and general exercises in a group setting for the remainder of their stay. Pre- and post- values of the listed outcome measures would be taken and analyzed.

The purpose of this fellowship is to determine if, through an educational and exercise class setting, improvements can be made in women with UI in an acute rehab hospital. Also, surveys will be used to see if patients find this type of intervention satisfactory and appropriate in this level of care. Another outcome of this fellowship will be to expand this intervention to other inpatient units and day rehab sites in the RIC system.

Specific Aim #1: To determine if women with urinary incontinence in an acute care rehab setting are satisfied with a group setting to treat UI Hypothesis 1: Women with urinary incontinence in an acute care rehab setting will find a group educational and exercise class appropriate for an acute care rehab hospital setting.

Specific Aim #2: To determine if women with urinary incontinence in an acute rehab setting feel the group setting of educational class of lecture and video and exercise class was effective in reducing the amount or severity of UI Hypothesis 2: Women with urinary incontinence in an acute care rehab setting will find a group educational (lecture and video) and exercise class effective in reducing the amount or severity of UI Specific Aim #3: To determine if women's quality of life improves with treating incontinence in an inpatient rehab setting Hypothesis 3: Quality of life will improve for women with urinary incontinence treated through group educational and exercise classes in an acute care rehab setting.

Methods This is a prospective pilot study of 15 women who have been admitted to the Rehab Institute of Chicago. There will not be a control group, and all 15 women will be in the intervention group. Patients will be selected from the 4th floor inpatient unit. Diagnoses will include women with orthopedic injuries, spinal surgeries, s/p surgical procedures, and general debility due to hospitalizations. All types of incontinence will be included in the study. UI will be defined as having an episode of loss of urine in the last 3 months.

1. Study participants will be recruited from the therapy (PT and OT), nursing, and medical staff on the 4th floor of the Rehabilitation Institute of Chicago by patient report during initial assessment/evaluations.
2. Investigator will determine if subject fits inclusion criteria for study by checking the medical record and subjective interview.
3. Participants will be recruited for a period of 8 months with the expectation to enroll 15 women.
4. The women who consent to participate in the study will be given a set of questionnaires at the time of consent and asked to complete by the next session.
5. Consenting patient will undergo an internal and external pelvic floor muscle examination. These procedures will be performed by the investigator.
6. If upon evaluation, the patient can perform the pelvic floor muscle contraction, she will then be enrolled in both an educational class and a pelvic floor exercise class. If extra time is needed for the patient to improve the contraction, the patient will receive more 1:1 time before being enrolled in the exercise class.
7. The educational class will focus on the anatomy of the pelvic floor, physiology of urination, urinary incontinence, behavioral modifications in bladder training, dietary impact on bladder function, and performance of pelvic floor muscle exercises. The exercise class will have an emphasis on pelvic floor exercises, core exercises, and general body conditioning.
8. An external and internal pelvic floor muscle examination will be performed after the intervention, prior to discharge to next level of care.
9. All intervention will be performed while the patient is in the hospital, and no follow-up visits will be required.
10. Participants will not be compensated for this study.

Recruitment

1. Staff nurses, resident physicians, attending physicians, nurse practitioners, physical or occupational therapists will inform investigator of any patient self-reports of incontinence by women admitted to the 4th floor nursing unit during initial evaluations or any other time during their stay.
2. The staff member will explain the study to the woman, and she will be asked if the study investigator could come and discuss the possibility of enrolling in this study.
3. The investigator will approach every woman referred to the study and will explain the study in more detail. Participants will be asked to sign the consent form if they agree to participate and allow collection of personal health information. Ample time will be allowed for reading and answering any questions.
4. After consent if gathered, the investigator will determine if the subject fits all inclusion/exclusion criteria.
5. Subject will be notified of investigators findings within 1 day of talking with the investigator for confirmation or exclusion of enrollment.

Analysis Following HIPPA guidelines, patient identifiable data will be coded to protect each patient's identity. The data obtained from the patients will be entered onto electronic teleforms and imported into the database. This is an RIC secure server where access will only be given to project staff. We are familiar with using this technology on other studies. It is efficient to complete in clinical setting and minimize data entry errors. The data will be used to describe patient characteristics and trends in findings.

We will run descriptive analyses to characterize the patients in the study. We will report the percent of patients who indicate they were satisfied with the program. We will compare pre-program and post-program outcomes using t-tests. Outcomes include: the frequency and severity of incontinence, quality of life, satisfaction with intervention, and FIM bladder score. Analyses will be conducted using SPSS version 20.

Outcome Measures Frequency and severity of Incontinence: We will be measuring this concept using the FIM data from the patient's medical chart to note the number of accidents reported in a 24 hour time frame. The severity of incontinence will be measured with the Sandvick's severity index, a valid measure to score the severity of urinary incontinence in women.

Quality of Life: The quality of life of these subjects will be tested using the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) Satisfaction: A satisfaction survey developed by the Principal Investigator will be used to understand the subject's satisfaction with the program.

Data Collection Time points Data will be collected at 2 separate time points. Data will be collected initially upon consent to the study and then again prior to subject discharge to the next level of care.

Data Collection Format Personal Health Information will be collected by the investigator through review of the subject's medical chart and subjective interview after consent to participate is received. Participants will be given paper copies of the survey questionnaires to complete and the investigator will collect the surveys. The results of the surveys and physical examinations will be entered onto an Excel spreadsheet by study personnel. All data will be stored on a password protected file in a RIC secure server with access only to project staff. No names will be included in the data files, only study identification numbers. The study identification numbers will be tracked in a separate data folder on the same secure network, also password protected. A detailed description of data to be collected follows.

.

Evaluation/Assessment:

Outcomes will consist of patient responses to standardized and non-standardized questionnaires and physical examination. In addition, we will collect relevant demographic data and medical utilization data to describe the study population.

Subjective interviews will be given to understand the specifics of each subject's urinary incontinence and previous treatments. A satisfaction survey will be developed by the principal investigator and given to subjects at the end of their enrollment. The purpose of the survey will be to determine if the information was understood and if the patient was satisfied with the type of interventions. The International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) will be used to look at quality of life issues with the participants before and after the intervention. The ICIQ-SF has been proven to show widespread applicability as an outcome measure in patients with incontinence. Admission FIM and discharge FIM score for the bladder management will be collected to address if the intervention was successful in decreasing the number of accidents/episodes of incontinence per day. All objective findings will follow the Laycock PERFECT Scale and ICS guidelines to standardize the terminology.

Tests and Measures:

The investigator will perform an external and internal pelvic floor muscle examination. This will include a sensory screen to external pelvic region, anal wink reflex, and external observation of perineal body mobility. Internally, the investigator will assess tone in pelvic floor musculature, and muscle strength will be assessed using the Modified Oxford scale and Laycock PERFECT scale.

Baseline and post-intervention ICIQ-SF and FIM scores will be compared using a one sample t-test (if normally distributed) or the Wilcoxon-Mann-Whitney test (if data are not normally distributed).

Physical Examination Procedures:

Internal Muscuoloskeletal Tests and Measures: During all procedures, unless otherwise noted, the patient will be disrobed below the waist and allowed to wear her choosing above the waist.

1. Internal assessment of pelvic floor muscle function: The examiner observes the movement of the patient's perineum with the patient in the supine position with legs spread or in the dorsal lithotomy position; approximate time for testing 2 minutes, graded as present or absent

   1. voluntary contraction: moves ventrally and cranially during contraction
   2. voluntary relaxation: able to relax on demand, descends from ventral position
   3. involuntary contraction: takes place preceding increase in abdominal pressure
   4. involuntary relaxation: takes place when straining as in defecation
2. Modified Oxford scale: The examiner inserts a finger into the patient's vagina to perform a manual muscle test of right and left pelvic floor muscles with the patient in the supine or dorsal lithotomy position using the modified Oxford scale ; approximate time for testing 3 minutes. The patient is instructed to contract her pelvic floor muscles.

   1. 0/5 = no discernible contraction of muscles
   2. 1/5 = flicker or pulsation is felt, no discernible lifting or tightening
   3. 2/5 = weak contraction, no discernible lifting or tightening
   4. 3/5 = moderate, some lifting of the posterior wall and some tightening around the examiner's finger, contraction is visible
   5. 4/5 = good, elevation of the vaginal wall is felt against resistance, drawing in of the perineum is felt, able to hold for 5 or more seconds
   6. 5/5 = strong resistance is felt; if two fingers are inserted, fingers will be approximated, able to hold for with 10 second hold
3. Laycock PERFECT scale. Approximate time for testing is 10 minutes

   1. P=Use modified Oxford scale and ICS guidelines
   2. E=List number of seconds contraction is held
   3. R=List number of repetitions contraction is hel
   4. F=list number of contractions that can be performed in 10 seconds
   5. E=elevation of posterior vaginal wall toward pubic bone (absent or present)
   6. C=Co-contraction of the deep abdominal muscles (absent or present)
   7. T=Timing-involuntary pelvic floor muscle contraction (absent or present)
4. Pelvic floor palpation exam: The patient is disrobed from the waist down and is lying supine with hips and knees flexed. The examiner inserts a finger into the patient's vagina and performs manual palpation of pelvic floor and obturator internus musculature for tenderness. Approximate time for testing 5 minutes.

   a. Right and left superficial genital muscles i. Anterior ii. Perineal body iii. posterior b. Right and left levator ani c. Right and left obturator internus

Personal Health Information to be collected The personal health information items that will be collected will include

1. Name
2. Date of birth
3. Age
4. Medical Record Number
5. Number of previous pregnancies
6. Number of previous deliveries
7. Types of previous deliveries
8. Dates of deliveries
9. Instrumentation during delivery
10. Previous gynecological/abdominal surgeries
11. Previous/current pelvic radiation
12. Current medications
13. History or neurological disease
14. History of urinary or fecal incontinence
15. Other treatments for urinary incontinence
16. Length of incontinence (time since onset)
17. Race
18. Income Level
19. Highest Level of Education
20. Payer
21. History of back pain
22. History of and type of prior physical therapy for pelvic floor rehab for UI

Impact and Significance Urinary incontinence is a very prevalent problem in women, even those who are admitted to inpatient rehab units. Previous studies on treating UI have been done on community dwelling women, not those that are in a hospital setting. The research has shown that there is both a need and want to treat this condition in an inpatient hospital. Interventions with physical therapy and behavioral modifications have been proven to be the best first line of treating this condition so should be tested in this patient population. Improvements could be made in the subjects' severity of incontinence, quality of life, self-efficacy, and possible discharge destination. This study will also be of benefit to the Rehab Institute of Chicago by bringing urinary incontinence to the forefront of the rehab team and improve the process and techniques in which it is managed.

ELIGIBILITY:
Inclusion Criteria:

Inclusion includes English-speaking women over the age of 18 who have been admitted to the Rehabilitation Institute of Chicago with reports of urinary incontinence in the past 3 months. Those who report "yes" to the screening questions who fit the above criteria will be screened by the principal investigator to ensure they fall into the criteria.

Exclusion Criteria:

Non-English speaking women under the age of 18, or those that do not give consent to participate in the study will not be enrolled. Also excluded will be any woman who has any chance of being pregnant or having an active urinary tract infection. No women with active infection lesions, unknown vaginal bleeding or those who have never had any kind of pelvic examination will be included in the study. Other exclusion criteria include women with a neurogenic bladder or admission FIM scores on sections Comprehension and Memory of below 4. Women with reports of significant pelvic pain or recent pelvic surgery or radiation or post-partum in last 6 months will be excluded.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of urinary incontinent episodes | per day

SECONDARY OUTCOMES:
Urinary incontinence severity | participants will be followed for the duration of their hospital stay, an average of 2 weeks
  Sandvick Severity Scale
ICIQ-SF | participants will be followed for the duration of their hospital stay, average of 2 weeks
  quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Laura Pickering, PT, Study Director — Shirley Ryan AbilityLab